CLINICAL TRIAL: NCT06270069
Title: Responsiveness and Minimal Important Change of Two Measures of Pain Intensity in People With Low Back Pain
Status: Not yet recruiting | Type: Observational
Sponsor: International Institute of Behavioral Medicines (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-001
Record Dates: First submitted 2024-02-05; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Excercise-based therapy — An individual 60-min motor training sessions twice a week for eight-week outpatient program, that included exercises aimed at improving postural control, strengthening and stabilizing the back muscles, and stretching

SUMMARY:
This is an observational study aimed at evaluating the responsiveness and minimal important change of two measures of pain intensity in people with low back pain. It consists of a battery of self-administered questionnaires which will be given to individuals with low back pain to complete before and after a rehabilitation treatment. Relationships among the different outcome measures will be also evaluated.

DETAILED DESCRIPTION:
This is an observational study aimed at evaluating the responsiveness and minimal important change of two different graphical ways to assess pain intensity in people with low back pain.

Literature found out that low back pain intensity is commonly assessed by a numerical rating scale ranging from no pain to the worst imaginable pain, once presented to responders horizontally. A different way to assess pain intensity could be to answer a similar numerical rating scale if set vertically.

In Literature there are not studies which head-to-head evaluate the responsiveness and minimal important change of these two ways of assessing pain intensity due to low back pain.

Participants will also have to complete self-reported outcome measures of disability, catastrophizing, fear of movement and self-efficacy, and correlations among these tools and the above two different ways to evaluate pain intensity will be evaluated. Descriptive statistics will be presented by taking into account the socio-demographic characteristics of the sample under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Non specific low back pain
* Adult age
* Ability to understand the Italian language

Exclusion Criteria:

* Refuse to adhere to the study
* Definite causes of low back pain
* Central or peripheral neurological signs
* Systemic illness or psychiatric deficits
* Recent myocardial infarction, cerebrovascular events, or chronic lung or renal diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-speciﬁc low back pain is deﬁned as low back pain not attributable to a recognizable, known speciﬁc pathology (eg, infection, tumour, osteoporosis, lumbar spine fracture, structural deformity, inﬂammatory disorder,radicular syndrome, or cauda equina syndrome).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
NRS | Immediately before the rehab treatment starts and immediately after the intervention
  Numerical Rating Scale; score 0-10 with higher estimates indicating higher levels of pain intensity (horizontal line)
Gauge of pain | Immediately before the rehab treatment starts and immediately after the intervention
  Numerical Rating Scale; score -5/+5 with lower estimates indicating higher levels of pain intensity (vertical line)

SECONDARY OUTCOMES:
ODI | Immediately before the rehab treatment starts and immediately after the intervention
  Oswestry Disability Index; score 0-50 with higher scores representing greater restriction to activities.
PCS | Immediately before the rehab treatment starts and immediately after the intervention
  Pain Catastrophizing Scale; score 0-52 with higher estimates showing higher catastrophizing
TSK | Immediately before the rehab treatment starts and immediately after the intervention
  Tampa Scale of Kinesiophobia; score 13-52 with higher estimates showing higher fear of movement
PSEQ | Immediately before the rehab treatment starts and immediately after the intervention
  Pain Self Efficacy Questionnaire; score 0-60 with higher estimates showing higher self-effficacy
GPE | Immediately after the intervention
  Global Perceived Effect (how much did the treatment received help your pain?); score -3 (it worsen a lot the things)/+3 (it helped a lot)

IPD SHARING:
Plan to Share IPD: No